CLINICAL TRIAL: NCT04171336
Title: Animal-assisted Group Therapy for Children and Adolescents Suffering From Chronic Primary Pain
Brief Title: Animal-assisted Therapy for Children and Adolescents With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAT for CPP
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Pragmatic trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Animal-assisted group therapy (Experimental)
  Interventions: Behavioral: Animal-assisted therapy

INTERVENTIONS:
Behavioral: Animal-assisted therapy — Six sessions of animal-assisted intervention for children and adolescents, group format. The sessions will focus on psycho-education on pain, mindfulness, defocusing, getting active, and resources. Additionally, the intervention includes two family visits.

SUMMARY:
Chronic pain is highly prevalent in children and adolescents, up to one in four children will develop pain that persists or recurs for three or more months. Chronic pain is not only linked to significant psychological, physical, and social concerns for affected children and their families, but also places an enormous burden on healthcare systems - in the United States, chronic pain costs around $19.5 billion dollars each year and ranks among the most expensive pediatric health problems. Chronic pain significantly decreases quality of life and is associated with numerous missing days at school or at work.

Several interventions exist, however, for some, the risk-benefit profile is not favorable, or the effect sizes are small and the clinical effect can be questioned. In general, a multidisciplinary approach that includes medical, psychological, and physiological aspects has been shown to be most promising in the treatment of chronic pain in children and adolescents.

Clinical impressions suggest that an Animal-assisted Therapy (AAT) intervention could be promising, but to the best of our knowledge, this is the first study to investigate the effectiveness of an AAT intervention for children and adolescents with chronic pain. With this pragmatic trials investigators aim to investigate the pre- and post-intervention differences in pain levels, levels of emotional distress, and quality of life within participants with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 8-15 years
* Suffering from chronic pain (i.e., persistent or recurrent pain for 3 or more months, associated with significant emotional distress or functional limitations)
* Willing to work with therapy animals
* Fluent in German
* Willingness to participate

Exclusion Criteria:

* children younger than 7 years or adolescents older than 16 years of age
* Acute pain
* Allergy to animals Aversion against animals

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
Pain Intensity assessed by Visual Analogue Scale | 12 weeks
  Self-reported pain intensity scored on a 0-10 scale, reported before and after each session. Higher scores indicate higher pain intensity.
Pain Severity assessed by Visual Analogue Scale | 6 weeks
  Self-reported pain severity scored on a 0-10 scale, reported before and after each session. Higher scores indicate higher pain severity.
Pain Interference assessed by Visual Analogue Scale | 6 weeks
  Self-reported pain interference scored on a 0-10 scale, reported before and after each session. Higher scores indicate more pain interference.
Pain Acceptance assessed by Visual Analogue Scale | 6 weeks
  Self-reported pain acceptance scored on a 0-10 scale, reported before and after each session. Higher scores indicate more pain acceptance.
Pain Defocussing assessed by Visual Analogue Scale | 6 weeks
  Self-reported pain defocussing scored on a 0-10 scale, reported before and after each session. Higher scores indicate more pain defocussing.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Koechlin, PhD, Principal Investigator — Faculty of Psychology, University of Basel, Switzerland; Cosima Locher, PhD, Principal Investigator — Faculty of Psychology, University of Basel, Switzerland; Jens Gaab, Prof Dr, Principal Investigator — Faculty of Psychology, University of Basel, Switzerland
Locations (1):
- Faculty of Psychology, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Locher C, Petignat M, Wagner C, Hediger K, Roth B, Gaab J, Koechlin H. Animal-Assisted Psychotherapy for Pediatric Chronic Pain: Case Series of an Open Pilot Study to Test Initial Feasibility and Potential Efficacy. J Pain Res. 2023 May 29;16:1799-1811. doi: 10.2147/JPR.S394270. eCollection 2023. PMID 37273273